CLINICAL TRIAL: NCT04682002
Title: Low-back Pain During Pregnancy and Its Psycho-social Implications. The Role of the Osteopathic Manipulative Treatment Within Its Multi-disciplinary Management. A Randomised Controlled Study
Brief Title: Low-back Pain During Pregnancy and Its Psycho-social Implications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Come Collaboration (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COME-02-20
Record Dates: First submitted 2020-12-15; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Pregnancy Related; Low Back Pain; Pelvic Girdle Pain
Keywords: osteopathic manipulative treatment; pregnancy; pain; low back pain; pelvic girdle pain; psychological factors
MeSH Terms: conditions — Low Back Pain; Pelvic Girdle Pain; Pain | interventions — Manipulation, Osteopathic; Mindfulness; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT + multidisciplinary path (Experimental): Patients in the experimental group will follow the obstetrician's and multidisciplinary path which provides osteopathic treatments, mindfulness, yoga, clinical nutrition, coaching and usual obstetric care.
  Interventions: Other: Osteopathic manipulative treatment; Other: Mindfulness; Other: Yoga; Other: Clinical nutrition; Other: Coaching
- Usual care (Other): Patients in control group will continue the routine obstetrical care as established by international guidelines
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Osteopathic manipulative treatment — OMT will be used to treat pregnancy women after having performed a manual osteopathic assessment. The first osteopathic evaluation is carried out during the 12th week, with the possibility to undertake a personalized treatment built on the needs of the single patient; the chosen techniques are based on the collected data by the operator. A "black-box" type of treatment is undertaken.
  Arms: OMT + multidisciplinary path
Other: Usual care — Administration of routine care based on international guidelines
  Arms: Usual care
Other: Mindfulness — Mindfulness group weekly meetings. Mindfulness practices consist of cognitive and behavioral treatments for depression and anxiety, including mindfulness-based stress reduction and mindfulness-based cognitive therapy.
  Arms: OMT + multidisciplinary path
Other: Yoga — Weekly yoga group meetings. Yoga is a mind-body practice that encompasses a system of postures, deep breathing, and meditation. In this context, yoga practice is adapted to pregnancy with the aim of benefit women who suffer from anxiety, depression, stress, low back pain, and sleep disturbances.
  Arms: OMT + multidisciplinary path
Other: Clinical nutrition — Nutritional advice to all women participating in the study at 12 weeks of pregnancy, with the possibility of starting an individualized path.
  Arms: OMT + multidisciplinary path
Other: Coaching — There will be five personalized coaching sessions during the pregnancy.
  Arms: OMT + multidisciplinary path

SUMMARY:
Pregnancy-related pelvic girdle pain (PPP) and pregnancy-related lumbar pain (PLBP) are two distinct symptoms, which can occur together as lumbar-pelvic pain.The primary objective is to measure the impact of osteopathic manipulative treatment on pregnancy-related lumbar and pelvic pain. The secondary objective is to study the interaction between pain and psycho-social factors during the gestational period.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-44
* Primiparae
* Single pregnancy
* Spontaneous pregnancy - fisiological pregnancy
* pregnancy >= 12 weeks
* low-back pain (between the 12th rib and the lumbo-pelvic region) and/or pelvic (in the pubic region and/or in one or both of the sacro-iliac joint and/or of the gluteal region) non specific
* consent to treatment
* absence of linguistic barriers

Exclusion Criteria:

* Women aged <18 o >44
* Pathological pregnancy, twins
* Metabolic pathologies
* Obstetrician's emergencies
* Pre-term birth
* Specific lumbar and/or pelvic pain - Genetics disorders
* Major congenital anomalies
* Absence of consent to treatment
* Presence of linguistic barriers

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in VAS at 6 months | 6 months
  Change from Visual Analogue Scale (VAS) of pain at 6 months. VAS values range from 0-10, where 10 means highest pain and 0 no pain
Change in ODI at 6 months | 6 months
  Change from Oswestry disability index 2.1° - Italian version (ODI) of the score at 6 months. The ODI represents a ten 6-point questionnaire. The first section rates the intensity of pain and the remaining ones cover the disabling effect of pain on typical daily activities: personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and travelling. Each item ranges from 0 to 5 and the sum of the 10 scores is expressed as a percentage of the maximum scores, varying from 0 (no disability) to 100 (maximum disability)
Change in PMI at 6 months | 6 months
  Change from Pregnancy mobility index (PMI) of the score at 6 months. PMI is a self-report questionnaire to assess mobility in relation to back and pelvic girdle pain. The PMI consists of three scales: daily mobility in the house, household activities and mobility outdoors. Every item has a score option from 0-3 (respectively 'no problems performing this task', 'some effort performing this task', 'much effort performing this task', 'performing this task is impossible or only possible with the aid of others'), which was transformed to a 0-100 scale. Each domain score is the mean of all included items.
Change in PGQ at 6 months | 6 months
  Change from Pelvic-girdle pain questionnaire (PGQ) of the score at 6 months. The PGQ is a condition-specific, patient-reported outcome measure designed to measure pregnancy-related back pain and pelvic girdle pain for use both during pregnancy and postpartum in research and clinical practice. The questionnaire includes items relating to 2 scales (activity/ participation and body functions [symptoms]). Self-report questionnaire of 20 activity items and 5 symptom items scored on a 4-point response scale. Each question is scored from 'Not at all' (0) to 'To a large extent' (3). Questions on the activity sub-scale range from difficulty with dressing, climbing stairs, doing housework, rolling in bed to pushing a shopping cart. Item scores are summed and transformed to yield a score of 0 to 100, where 100 is the worst possible score.

SECONDARY OUTCOMES:
Change in PWB at 6 months | 6 months
  Change from Ryff's Psychological Well-Being Scales (PWB) of the score at 6 months. Ryff, the 42-item Psychological Wellbeing (PWB) Scale measures six aspects of wellbeing and happiness: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Respondents rate how strongly they agree or disagree with 42 statements using a 7-point scale (1 = strongly agree; 7 = strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Niccolò Giovanni, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico

IPD SHARING:
Plan to Share IPD: No
available upon request